CLINICAL TRIAL: NCT01834742
Title: Pharmacodynamic Evaluation of Stool Output Following Oral Administration of Various Low Volume PEG3350-based Gut Cleansing Solutions Using the Split Dose Intake in Healthy Subjects
Acronym: OUT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norgine (Industry)
Collaborators: Pierrel Research Europe GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NER1006-01/2011 (OUT)
Record Dates: First submitted 2013-04-15; First posted 2013-04-18 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Colorectal Cancer
Keywords: Moviprep; PEG3350; Laxative; Stool Output
MeSH Terms: conditions — Colorectal Neoplasms | interventions — MoviPrep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Part A, arm 1 (Experimental): Evening dose 1 plus fixed morning dose
  Interventions: Drug: NER1006
- Part A, arm 2 (Experimental): Evening dose 2 plus fixed morninf does
  Interventions: Drug: NER1006
- Part A, arm 3 (Experimental): Evening dose 3 plus fixed morning dose
  Interventions: Drug: NER1006
- Part A, arm 4 (Active Comparator): Moviprep
  Interventions: Drug: Moviprep
- Part B, arm 1 (Experimental): Fixed evening dose plus morning dose 1
  Interventions: Drug: NER1006
- Part B, arm 2 (Experimental): Fixed evening dose plus morning dose 2
  Interventions: Drug: NER1006
- Part B, arm 3 (Experimental): Fixed evening dose plus morning dose 3
  Interventions: Drug: NER1006
- Part B, arm 4 (Experimental): Fixed evening dose plus alternative morning dose
  Interventions: Drug: NER1006

INTERVENTIONS:
Drug: NER1006 — Single evening dose of 750mL solution containing 100g PEG3350 plus 6g sodium sulphate. Single morning dose containing 40g PEG3350, 33.9g sodium ascorbate, 20.1g ascorbic acid.
  Arms: Part A, arm 1
Drug: NER1006 — Single evening dose of 750mL solution containing 100g PEG3350 plus 9g sodium sulphate. Single morning dose containing 40g PEG3350, 33.9g sodium ascorbate, 20.1g ascorbic acid.
  Arms: Part A, arm 2
Drug: NER1006 — Single evening dose of 750mL solution containing 75g PEG3350 plus 5.6g sodium sulphate. Single morning dose containing 40g PEG3350, 33.9g sodium ascorbate, 20.1g ascorbic acid.
  Arms: Part A, arm 3
Drug: Moviprep — Reconstituted and administered in accordance with recommended split dose intake: one litre in the evening, one litre the following morning.
  Arms: Part A, arm 4
Drug: NER1006 — Single evening dose containing formulation selected from Part A of study. Single morning dose containing 40g PEG3350 and 56.6g sodium ascorbate.
  Arms: Part B, arm 1
Drug: NER1006 — Single evening dose containing formulation selected from Part A of study. Single morning dose containing 40g PEG3350, 33.9g sodium ascorbate and 21.4g magnesium ascorbate.
  Arms: Part B, arm 2
Drug: NER1006 — Single evening dose containing formulation selected from Part A of study. Single morning dose containing 40g PEG3350, 6g sodium sulphate and 33.9g sodium ascorbate.
  Arms: Part B, arm 3
Drug: NER1006 — Single evening dose containing formulation selected from Part A of study. Single morning dose containing 29g PEG3350 and 4.8g sulphate and 23.3g ascorbic acid.
  Arms: Part B, arm 4

SUMMARY:
This study is to investigate the effect of various modified low volume polyethylene glycol (PEG) 3350 and ascorbic acid/ascorbate (PEG+ASC)-based gut cleansing solutions on stool output in healthy subjects. In addition, the study is to assess and compare the safety and tolerance of the modified PEG+ASC formulations following oral administration with the safety profile of MOVIPREP®.

ELIGIBILITY:
Inclusion Criteria:

1. The subject's written informed consent must be obtained prior to inclusion.
2. Healthy subjects with an age of 18 to 45 years.
3. Healthy subjects need to be without any history of clinical significant gastrointestinal symptoms by clinical judgement and without the presence of acute abdominal discomfort or symptoms.
4. Females must be surgically sterile, practicing true sexual abstinence or using an acceptable form of effective contraception throughout the study from the following list: contraceptive implants, injectables, oral contraceptives, intrauterine system (IUS), some intrauterine devices (IUDs), vasectomised partner or barrier method (condom or occlusive cap) with spermicidal foam/gel/film/cream/suppository. Hormonal and IUD methods of contraception must be established for a period of 3 months prior to dosing and cannot be changed or altered during the study. All females must have a negative pregnancy test at screening and check-in.
5. Willing, able and competent to complete the entire procedure and to comply with study instructions.

Exclusion Criteria:

1. Use of laxatives in the last 12 months or colon motility altering drugs in the last 6 months.
2. Use of any prescription or over-the-counter (OTC) medication within 4 weeks prior to the first dose of investigational drug (excluding hormonal contraception, and occasional use of nonsteroidal anti-inflammatory drugs [NSAID], acetaminophen or metamizole).
3. Donation or loss of 500 mL or more of blood within 8 weeks prior to the first dose of investigational drug.
4. Any evidence of the history or presence of organic or functional gastrointestinal conditions (e.g. chronic constipation, irritable bowel syndrome [IBS], inflammatory bowel disease [IBD]).
5. Exhibiting relevant abnormal gastrointestinal motility according to clinical judgement in the past or now.
6. History or presence of any clinically significant acute illness within the 4 weeks prior to the first dose of investigational drug based on clinical judgement at screening and check-in evaluation.
7. Known glucose-6-phosphatase dehydrogenase deficiency.
8. Known phenylketonuria.
9. History or evidence of any clinical significant systemic cardiovascular, hepatic, pulmonal, neurological, metabolic and/or renal organ dysfunction.
10. History of clinically significant drug allergy; history of atopic allergy (asthma, urticaria, eczematous dermatitis), known hypersensitivity to polyethylene glycols and/or ascorbic acid.
11. History or evidence of any clinically relevant electrocardiogram (ECG) abnormalities and hypertension.
12. Evidence of dehydration.
13. Any evidence for abnormal sodium or potassium levels or clinically significant other electrolyte disturbances.
14. Females who are pregnant, having a positive pregnancy test at screening and/or admission to unit or planning a pregnancy. Females not using reliable methods of birth control.
15. Clinically relevant findings on physical examination based on Investigator's judgement.
16. Clinically relevant deviations of laboratory parameters from reference ranges at screening or check-in evaluation.
17. Positive serology for chronic viral hepatitis or human immunodeficiency virus (HIV) at screening.
18. History of drug or alcohol abuse within the 12 months prior to dosing or evidence of such abuse as indicated by the laboratory assays conducted during the screening or check-in evaluations.
19. Subjects who are unwilling to comply with the provisions of the study protocol.
20. Concurrent participation in an investigational drug study or participation within 3 month of study entry.
21. Subject has a condition or is in a situation, which in the Investigators opinion may put the subject at significant risk, may confound the study results, or may interfere significantly.
22. Previous participation in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 161 (Actual)
Dates: Start 2011-04; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Primary Variable | 36 Hours
  Stool weight output generated from the start of intake for the following 24 hours.

SECONDARY OUTCOMES:
PEG3350 concentration | 96 Hours
  Concentration of PEG3350 in blood, urine and faeces.
Sulphate concentration | 96 hours
  Concentration of PEG3350 in blood, urine and faeces.
Ascorbic acid concentration | 96 hours
  Concentration of ascorbic acid in blood, urine and faeces.
Electrolytes concentration | 96 hours
  Concentration of electrolytes in blood, urine and faeces.
Safety profile | 96 hours
  Spontaneouly reported adverse events will be recorded throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Rodica Cinca, MD, Principal Investigator — Pierrel Research
Locations (1):
- Pierrel Research HP-RO-SRL, Timișoara, Romania